CLINICAL TRIAL: NCT01669824
Title: Tolerability, Compliance and Indications of Aspirin Protect 100 mg in Longterm Use (12 Months) Under Everyday's Conditions - Data Collection With Questionnaires Handed Out in Pharmacies to Aspirin Protect 100 mg Consumers
Brief Title: Pharmacy Based Pharmacoepidemiological Observational Study With Aspirin Protect 100 mg
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Country Medical Director, Bayer Vital GmbH
Other Study IDs: 12557; MUE 053 (Other: Company internal)
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2012-08

CONDITIONS: Aspirin; Drug Safety; Effects, Longterm
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465)

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin, BAYE4465) — Aspirin protect (enteric coated aspirin) 100 mg/single dose/day as long-term medication

SUMMARY:
In this non-interventional one year study, data about overall and particularly gastrointestinal tolerability, indications, cardiovascular risk factors and compliance are collected by basic questionnaires, which are handed out by pharmacists to patients who acquire (in Germany no prescription is needed) Rx (Prescription) or OTC (Over-The-counter) Aspirin protect (enteric coated aspirin) 100 mg and are willing to participate in the study. After 3, 6, 9 and 12 months follow-up questionnaires are sent out. Aim of the study is to get information about safety, usage and compliance under everyday's conditions, because in Germany low-dose aspirin is an OTC product with Rx indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients who buy Aspirin protect 100 mg in a pharmacy and are willing to participate in the study.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who buy Aspirin protect 100 mg with or without prescription in German pharmacies and who are willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 4235 (Actual)
Dates: Start 2007-08; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Overall and gastrointestinal tolerability assessed by questionnaire | After 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Germany